CLINICAL TRIAL: NCT06925178
Title: Multi-Modality Imaging Standard Cohort Of Cerebrovascular Disease
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zi-Xiao Li, Professor, Beijing Tiantan Hospital
Other Study IDs: HX-B-2024061
Record Dates: First submitted 2024-11-20; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-11

CONDITIONS: Cerebrovascular Disease
Keywords: stroke; progonosis; imaging; cognitive disorder
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to establish a multi-center and multi-modality imaging standard cohort of cerebrovascular disease, analyze the potential mechanisms affecting the prognosis of cerebrovascular disease based on a variety of imaging methods, and explore potential therapeutic targets.

DETAILED DESCRIPTION:
Cerebrovascular diseases are major diseases that pose a serious threat to human health and life, and have become the leading cause of death from disease among Chinese residents. Despite the best medical or surgical treatment options, many patients still suffer from functional disabilities, imposing a heavy burden on families and society. Identifying the complex and delicate changes in brain neural activity, blood flow, oxygenation, and metabolism following the occurrence of cerebrovascular diseases can not only explore the potential mechanisms underlying poor functional prognosis, but also provide a scientific basis for targeted treatment strategies. This study is a consecutive, multicenter, prospective registration study that recruits approximately 800 patients with cerebrovascular diseases (both hemorrhagic and ischemic stroke) aged 18-80 years within 7 days of onset. The study collects baseline information and imaging data including head CT, MRI, TCD, fNIRS, and ophthalmic testing. The primary endpoint event was functional outcome 3 months (mRS score). Secondary outcomes were in-hospital complications (including stroke progression, recurrence, and mortality), cognitive disorder, functional outcomes, recurrent stroke, new vascular events, and all-cause death at 3, 6 and 12 months .

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old;
* Onset of symptoms within 7 days;
* Clinical diagnosis of cerebrovascular disease (ischemic stroke or hemorrhagic stroke) confirmed by head imaging (CT or MRI);
* Signed informed consent form.

Exclusion Criteria:

* Diagnosed with non-cerebrovascular diseases (such as central nervous system infections, epilepsy, and metabolic encephalopathy);
* Patients with contraindications to multimodal CT or MRI, functional near-infrared imaging, or those who cannot cooperate to complete the relevant examinations;
* Patients with a life expectancy of less than 3 months or those who cannot complete the study follow-up due to other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-80 years old with acute cerebrovascular disease (hemorrhagic or ischemic stroke) within 7 days of onset； healthy adults.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of unfavorable functional outcome | 3 month after enrollment
  Unfavorable functional outcome is defined as mRS Score 2-5. mRS is an efficient, reliable and simple scale to assess the recovery of neurological function and disability after stroke. The high score indicates the poor neurological recovery. The minimum score (0) means no symptoms at all. The maximum (6) means death.

SECONDARY OUTCOMES:
The incidence of in-hospital complications | duration of hospital stay（about 1 week）
  In-hospital complications (including stroke progression, recurrence, and mortality).
The incidence of unfavorable functional outcome | 6 and 12 months after enrollment
  Unfavorable functional outcome is defined as the modified Rankin Scale (mRS) Score 2-5. mRS is an efficient, reliable and simple scale to assess the recovery of neurological function and disability after stroke. The high score indicates the poor neurological recovery. The minimum score (0) means no symptoms at all. The maximum (6) means death.
The incidence of new vascular events | 3, 6 and 12 months after enrollment
  Including ischemic stroke, hemorrhagic stroke, myocardial infarction or vascular death.
The incidence of recurrent stroke | 3, 6 and 12 months after enrollment
  Stroke recurrence is defined as a new focal neurological impairment that was confirmed by neuroimaging, including both ischemic stroke and hemorrhagic stroke.
The incidence of all-cause death | 3, 6 and 12 months after enrollment
  An all-cause death is defined as a death from any cause.
The incidence of Cognitive impairment | 3, 6 and 12 months after enrollment
  Cognitive impairment is assessed using the MMSE and MOCA scales, with scores below 27 on the MMSE or below 26 on the MOCA indicating the presence of cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No